CLINICAL TRIAL: NCT03836196
Title: Optimizing the Management of High-risk and Unfavorable Intermediate-risk Disease: the Use of Advanced Imaging, Trans-perineal Mapping Biopsies, and Dual-strength Brachytherapy Sources to Minimize Radiation Dose to Normal Tissues
Brief Title: Optimizing Prostate Cancer Treatment in Men With Advanced Local Disease
Acronym: OPTiMAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: H18-01937
Record Dates: First submitted 2018-11-20; First posted 2019-02-11 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; PSMA PET/CT; multi-parametric MRI; multi-parametric TRUS; Transperineal mapping biopsy; LDR Brachytherapy; External Beam Radiation Treatment
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combined radiation treatment (Experimental): Combined low-dose-rate brachytherapy and external beam radiation therapy
  Interventions: Radiation: LDR Brachytherapy and External Beam Radiation Therapy

INTERVENTIONS:
Radiation: LDR Brachytherapy and External Beam Radiation Therapy — Low Dose Rate Brachytherapy (LDR-PB) and External Beam Radiation Therapy (EBRT)

SUMMARY:
Multi-modality therapy that includes a brachytherapy implant improves outcomes in locally advanced prostate cancer when compared to other radiation-based treatments, but is also associated with more adverse side effects. The goal of the OPTiMAL trial is to reduce these side effects by using advanced imaging and biopsy techniques to locate cancer and deliver precision radiation therapy, while not compromising the unprecedented high cure rates obtained for the brachytherapy arm of the Androgen Suppression Combined with Elective Nodal and Dose Escalated Radiation Therapy (ASCENDE-RT) randomized control trial.

Additionally, some applied research in genetics, pathology and medical imaging is included. Novel medical imaging methods, namely, multi-parametric magnetic resonance imaging (MRI), multi-parametric trans-rectal ultrasound (TRUS), prostate-specific membrane antigen (PSMA) positron emission tomography/computed tomography (PET/CT) are used for re-staging of prostate cancer. This is followed by trans-perineal biopsy to locate cancerous areas of the prostate with greater precision compared to conventional biopsy. Results from imaging are compared to those from biopsy to develop image-based cancer detection methods.

DETAILED DESCRIPTION:
Purpose:

The purpose of OPTiMAL is to combine new imaging and treatment methods to reduce the incidence and severity of the genito-urinary (GU) side effects associated with radiation-based, multimodality treatment for men with locally advanced prostate cancer (PCa). OPTiMAL was inspired by the highly successful Androgen Suppression Combined with Elective Nodal and Dose Escalated Radiation Therapy (ASCENDE-RT) randomized control trial, in which men who were randomized to a low-dose-rate brachytherapy (LDR-PB) boost experienced unprecedented high cure rates, but also had more side effects and a slightly greater decrease in quality-of-life (QoL) scores when compared to the standard arm which used a dose-escalated external beam (DE-EBRT) boost.

Hypothesis:

By allowing a higher radiation dose to the cancer while delivering lower dose to healthy tissue, more accurate cancer localization will result in a decrease in adverse effects and better QoL, when compared to the men in the experimental arm of ASCENDE-RT.

Justification:

About 1 in 4 newly diagnosed PCa patients will be found to have unfavorable disease , either National Comprehensive Cancer Network (NCCN) high-risk or intermediate-risk with multiple adverse features; such men carry a 40% to 80% chance of biochemical recurrence within 5 years of radical prostatectomy (RP) or conventional external beam radiation therapy (EBRT) alone. With some exceptions, such men generally require multi-modality treatment to provide the best chance of long-term disease-free survival.

In the ASCENDE-RT randomized control trial, led by investigators at BCCANCER, an LDR-PB boost established unprecedented new standards for biochemical (PSA) progression free survival (b-PFS); however, a higher incidence of adverse GU side effects was also observed. Despite the increase in adverse effects, most men were symptom-free at 5 years and more than 80% had minimal or no adverse effects left over from treatment.

Objectives:

Primary objective:

OPTiMAL is powered to determine if combining improved techniques for delivering combined pelvic EBRT and LDR-PB boost will lead to a reduction in grade 2 and above, physician-reported GU adverse effects when compared to the ASCENDE-RT trial while not compromising the high rates of biochemical progression free survival survival (b-PFS) observed in ASCENDE-RT.

Secondary Objectives:

1. Trans-perineal, template-guided mapping biopsy (TTMB) is the gold standard for locating the extent of intra-prostatic disease, but it is an invasive procedure. Therefore, another objective of this trial is to establish and investigate correlations between TTMB and multi-modality, multi-parametric imaging provided by trans-rectal ultrasound (TRUS), MRI and PET/CT.
2. To further develop the use of dual air kerma strength sources in a single LDR-PB implant, which the investigators have shown can improve the planning target volume (PTV) dose coverage while reducing dose to sensitive normal tissues.
3. Finally, the TTMB biopsy material will also be used to compare computer-based digital pathology to conventional pathology as read by human pathologists.

Research design:

Eligible patients will undergo a series of re-staging investigations, which includes multiple advanced imaging: PSMA PET/CT, Multi-parametric MRI and TRUS and trans-perineal biopsy. Re-staging will be used to determine which components of multi-modality therapy are appropriate for each individual patient.

Treatment includes a combination of 125 iodine LDR-PB, followed by EBRT. Based on the results from the re-staging phase and baseline patient diagnosis, in some cases androgen deprivation therapy will be prescribed for a total duration of at least one year with at least 6 months being neoadjuvant.

125 Iodine LDR-PB implant will be designed to deliver a minimum peripheral dose (MPD) of 100 Gy to the entire gland and a boost of 150-200 Gy either to the entire peripheral zone, or in cases with well-localized intra-prostatic disease on the basis of TTMB, to regions of known disease only. For all trial subjects the use of dual strength source may be used if their use results in superior coverage and/or protection of normal tissues

Shortly after the completion of the LDR-PB implant, all patients will receive supplemental pelvic EBRT using Volumetric Modulated Radiation Therapy (VMAT) intensity modulated radiation therapy (IMRT).

Statistical Analysis:

The study will include a total of 105 enrolled patients who will receive multi-parametric imaging and TTMB over 4 years. Based on the investigators' experience at the BCCANCER, it is estimated that 75 patients will receive focal LDR-PB boost.

Assuming that the 2-year cumulative incidence rate of grade 2 or above toxicity is similar to the DE-EBRT arm of the ASCENDE-RT trial (10%), a study exposing 75 subjects to focal LDR-PB boost is sufficient to demonstrate a cumulative incidence significantly lower than the 26% in the LDR-PB boost arm of ASCENDE-RT with 96% power based on a two-sided 95% confidence interval of the Kalbfleisch-Prentice incidence estimator. Enrolling 75 subjects over 4 years with 2 years of follow-up and assuming the 2-year rate of grade 3 or above toxicity is 3.4%, the 95% confidence interval for 2-year incidence will exclude 7.7% with more than 81% power.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically-proven prostate cancer
* Patients must meet either: a. National Comprehensive Cancer Network (NCCN) definition of high-risk disease or b. Intermediate-risk disease with at least 3 points using the following scale: One point each for clinical stage = T2b-c, iPSA >7 ng/mL, and Gleason grade group 2 (overall Gleason sum 3+4 =7), Two points for Gleason grade group 3 (overall Gleason sum 4+3 =7).
* Patients must have N0 M0 status on the basis of technetium bone scan and computed tomography (CT) scan of the pelvis

Exclusion Criteria:

* Those with pre-intervention prostate specific antigen (iPSA) above 100 ng/mL.
* Those who have received prior surgical treatment for prostate cancer including transurethral resection of the prostate (TURP), transurethral resection of the bladder neck (TURB), cryotherapy, laser ablation, or high frequency ultrasound (HIFU)
* Those with an estimated life expectancy of less than 5 years with an Eastern Cooperative Oncology Group (ECOG ) performance status above 0-2
* Those with prior radiation therapy to the pelvis.
* Those who have received androgen deprivation therapy (ADT) prior to registration.
* Contraindication to high-dose pelvic irradiation, Luteinizing hormone-releasing hormone (LHRH) agonists, or nonsteroidal antiandrogen therapy
* Those who are not able to participate in an MRI scan (i.e. significant renal impairment that would preclude the use of contrast agent, some patients with cardiac pacemaker, wires, or defibrillator; artificial heart valve; brain aneurysm clip; electrical stimulator for nerves or bones; ear or eye implant; implanted drug infusion pump; coil; catheter, or filter in any blood vessel. Some men with metallic prosthesis; shrapnel, bullets, or other metal fragments retained in the body)
* Those who are not able to participate in a PET/CT scan
* Cancer survivors who do not meet all three of the following criteria: a) The patient has undergone potentially curative therapy for all prior malignancies. b) There has been no evidence of recurrence for at least five years following potentially curative therapy. (For non-melanoma skin cancer the five-year requirement does not apply.) and c) The patient is considered by the treating physician to be at low risk of recurrence from prior malignancies.
* Those who are on anticoagulation therapy (blood thinners) and are unable stop this medication safely for at least 5 days.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2019-09-13 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Frequency of treatment-related GU adverse effects | Analysis to be done at median follow-up of 2 years
  Cumulative frequency of Physician-reported grade 2 and above GU adverse events (scored using a modified CTCAE - Common Terminology Criteria for Adverse Events- scale).

SECONDARY OUTCOMES:
Trans-perineal biopsy and imaging correlation | 2 years
  Correlations between trans-perineal biopsy and multi-modality, multi-parametric imaging provided by multi-parametric TRUS, multi-parametric MRI and PSMA PET/CT

CONTACTS AND LOCATIONS:
Overall Officials: Michael Peacock, MD, Principal Investigator — BCCANCER
Locations (1):
- BC Cancer - Vancouver, Vancouver, British Columbia, Canada